CLINICAL TRIAL: NCT05481944
Title: Metabolic Inflexibility of the Heart as a Predictor of Occurrence of Heart Failure in Patients With Type 2 Diabetes
Acronym: MET-INF-T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP190632
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; insulin therapy; metabolic inflexibility
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with insulinotherapy introduction (Active Comparator): Injected MRI
  Interventions: Diagnostic Test: MRI in patients
- Healthy volunteers (Sham Comparator): No injected MRI
  Interventions: Diagnostic Test: MRI in healthy volunteers

INTERVENTIONS:
Diagnostic Test: MRI in patients — Injected MRI
  Arms: Patients with insulinotherapy introduction
Diagnostic Test: MRI in healthy volunteers — non injected MRI
  Arms: Healthy volunteers

SUMMARY:
In the type 2 diabetic population, some patients are particularly at risk of developing early heart failure. Finding markers to identify these at-risk individuals is therefore an important scientific objective in order to avoid/delay the development of heart failure.

The protocol will be proposed to type 2 diabetic patients hospitalized for insulin therapy upon admission to the diabetology department and healthy volunteers.

DETAILED DESCRIPTION:
The objective of this study is to identify subjects at risk defined by the existence of an alteration in the maximal longitudinal contractility of the left ventricle by measuring myocardial deformation in magnetic resonance imaging (MRI) before (D1) and after (D15±3) an imposed metabolic change (insulin treatment and correction of hyperglycaemia) in a population with type 2 diabetes in primary prevention requiring the start of insulin therapy because of an imbalance in their diabetes (HbA1c ≥ 10%). To do so, patients and healthy volunteers will be matched on sex and age (+/- 5 years).

ELIGIBILITY:
Inclusion Criteria:

Patients

* Patient aged over 18 and under 75
* Type 2 diabetes treated with bitherapy for at least 6 months
* Unbalanced diabetes (HbA1c ≥ 10%)
* Indication for insulin therapy (introduction of a slow-acting insulin injection per day or adding rapid-acting insulins before meals in the event of a slow-acting or semi-acting insulin injection already present on admission)
* BMI < 40 kg/m2
* Cardiovascular examination without clinically significant abnormality
* LVEF > 50% (measured by echocardiography)
* Free from any acute intercurrent pathology for more than 10 days,
* Accept the constraints of the protocol and sign the informed and free consent
* Be affiliated to a French social security scheme or entitled

Healthy volunteers

* Be over 18 and under 75
* Have a BMI < 30 kg/m²
* Be asymptomatic
* Normal clinical examination
* Normal resting 12-lead ECG
* Normal biological balance (fasting blood glucose, HBA1c, ionogram, creatinine, NFS, BNP / pro-BNP, troponin)
* Accept the constraints of the protocol and sign the informed and free consent
* Be affiliated to a French social security scheme or entitled

Exclusion Criteria:

Patients

* Current or recent infections (< 10 days)
* Neoplastic disorders (except carcinoma in situ of the cervix or cutaneous epithelioma), haematological, cardiovascular (except controlled arterial hypertension), psychiatric, neurological, chronic respiratory failure
* Presence of renal insufficiency defined as an estimated glomerular filtration rate < 30mL/min/1.73m2 according to the MDRD formula
* Rhythm and/or conduction disorder not previously known and discovered during the 12-lead ECG performed at inclusion
* Known cardiovascular pathology (arteriopathy and/or cardiomyopathy)
* Contraindications to MRI with injection of gadolinium: claustrophobia, pacemaker, metallic foreign body, anxiety attack, nausea, vomiting, panic attack, vertigo, malaise without traumatic consequences, allergy to contrast products, renal failure defined by an estimated glomerular filtration rate < 30mL/min/1.73m2 according to the MDRD formula, diffusion of the contrast product during its infusion
* Contraindication for regadenoson injection: hypersensitivity to the active substance or to any of the excipients, second or third degree atrioventricular (AV) block or sinoatrial node dysfunction, unless these patients are carriers an operational pacemaker, unstable angina not stabilized by medical treatment, severe hypotension, decompensated heart failure
* Pregnant or breastfeeding women
* Persons deprived of their liberty by judicial decision or benefiting from legal protection (under guardianship or curatorship)
* Abuse of alcohol or narcotics
* Patient under AME (state medical aid)
* Participation in another interventional research involving the human person or being in the exclusion period at the end of a previous research involving the human person

Healthy volunteers

* Contraindications to MRI: claustrophobia, metallic foreign body, anxiety attack, nausea, vomiting, panic attack, vertigo, malaise without traumatic consequences
* Have kidney disease with GFR < 30 mL/min
* Known cardiac pathology
* Personal cardiovascular history
* Primary cardiomyopathy or familial congenital heart disease
* Being deprived of liberty or under legal protection (under guardianship or curatorship)
* Witness under AME (state medical aid)
* Participation in another interventional research involving the human person or being in the exclusion period at the end of a previous research involving the human person
* Pregnant or breastfeeding woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Left ventricular myocardial longitudinal strain measured by MRI (%) | 15 days
  Myocardial longitudinal strain measured by dynamic MRI images (%) throughtout feature tracking strategy

SECONDARY OUTCOMES:
Left ventricular myocardial radial strain measured by dynamic MRI images (%) throughtout feature tracking strategy | 15 days
Extracellualar volume (%) and collagene fraction (%) measured from MRI images | 15 days
Rest ratio in myocardial perfusion reserve calculated from rest and stress MRI images | 15 days
Measurement of early and late filling wave velocities (E, A) and myocardial longitudinal velocity (E') | 15 days
Myocardial triglycerides fraction measured from proton MR spectroscopy | 15 days
Epicardial fat volume measured from ECG gated Dixon MRI images | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio ANDREELLI, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission Nationale de l'Informatique et des Libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal